CLINICAL TRIAL: NCT04307940
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Compare the Analgesic Efficacy and Safety of Naproxen Sodium Tablets and Hydrocodone/Acetaminophen Tablets in Postsurgical Dental Pain
Brief Title: Study to Collect Information on How Well the Study Drug Naproxen Sodium Tablets Works Compared to Hydrocodone/Acetaminophen Tablets in Order to Relieve Pain in Participants Experiencing Moderate to Severe Pain After Having Their Wisdom Teeth Removed
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20536
Record Dates: First submitted 2020-03-05; First posted 2020-03-13 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pain
Keywords: Postsurgical Dental Pain
MeSH Terms: conditions — Pain | interventions — Naproxen; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Naproxen sodium (Experimental): After completion of the surgical teeth extractions, qualified participants will be randomized into one of three treatments with a 2:2:1 ratio. (Naproxen sodium=2, Hydrocodone/Acetaminophen=2, Placebo=1)
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031)
- Hydrocodone/Acetaminophen (Active Comparator): After completion of the surgical teeth extractions, qualified participants will be randomized into one of three treatments with a 2:2:1 ratio. (Naproxen sodium=2, Hydrocodone/Acetaminophen=2, Placebo=1)
  Interventions: Drug: Hydrocodone/Acetaminophen
- Placebo (Placebo Comparator): After completion of the surgical teeth extractions, qualified participants will be randomized into one of three treatments with a 2:2:1 ratio. (Naproxen sodium=2, Hydrocodone/Acetaminophen=2, Placebo=1)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen Sodium (Aleve, BAY117031) — 220 mg per tablet, two tablets (440 mg), intake a single dose orally.
  Arms: Naproxen sodium
Drug: Hydrocodone/Acetaminophen — 5/325 mg per tablet, two tablets (10/650 mg), intake a single dose orally.
  Arms: Hydrocodone/Acetaminophen
Drug: Placebo — two tablets, intake a single dose orally.
  Arms: Placebo

SUMMARY:
With this study researchers want to collect information on how long the pain relief lasts after a fixed dose of naproxen sodium or hydrocodone/acetaminophen or placebo (contains no medication) over 12 hours in subjects experiencing moderate to severe pain after having their wisdom teeth removed. Naproxen Sodium (Aleve®) is a drug that is used for the temporary relief of minor aches and pains.

Hydrocodone/Acetaminophen is a combination drug used to relieve moderate to severe pain. It contains an opioid (narcotic) pain reliever (hydrocodone) and a non-opioid pain reliever (acetaminophen).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male or female volunteers 18 to 40 years of age;
* Subjects will undergo surgical extraction of three or four third molars, two of which must be mandibular molars. Maxillary third molars may be removed regardless of impaction level. The mandibular extractions must have a trauma rating of mild or moderate and meet one of the following scenarios:

  * two full bony impactions
  * two partial bony impactions
  * one full bony impaction in combination with one partial bony impaction Supernumerary teeth present may also be removed at the discretion of the oral surgeon;
* Have not consumed alcoholic beverages, or foods and beverages containing caffeine (examples; coffee, tea, chocolate, and colas) after midnight prior to surgery and agree not to consume any of these foods or beverages throughout their stay at the study site;
* Use of only short-acting local anesthetic (e.g., mepivacaine or lidocaine) preoperatively, with or without a vasoconstrictor and nitrous oxide at the discretion of the Investigator;
* Have moderate to severe postoperative pain on the Categorical Pain Intensity Scale (a score of at least 2 on a 4 point scale) and a score of ≥ 5 on the 0-10 pain intensity NRS within 4.5 hours postsurgery;
* Ability to understand and follow study-related instructions;
* Be willing and able to participate in all scheduled visits, treatment plan, and trial procedures according to the clinical protocol;

Exclusion Criteria:

* History of hypersensitivity to naproxen sodium, hydrocodone/acetaminophen, ibuprofen, NSAIDS, aspirin, similar pharmacological agents, local anesthetics, rescue medication or components of the investigational products;
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including hypertension), hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years;
* Subjects with the following medical conditions may be eligible at the discretion of the investigator: ADHD on a stable dose regimen of methylphenidate/(dextro)amphetamine for at least 6 months; subjects with hypothyroidism on a stable dose of synthetic thyroid hormone for at least 6 months;
* Have received any form of treatment in the form of medication for depression in the past 6 months or any form of psychotropic agent (including selective serotonin uptake inhibitors [SSRI] but excluding ADHD medications described above) within the last 6 months;
* Use of any OTC or prescription medications with which the administration of naproxen, hydrocodone/acetaminophen, acetaminophen, ibuprofen, any other NSAID, (e.g., tramadol) or if a medication is contraindicated;
* Females who are planning to become pregnant, pregnant or lactating;
* Habituation to analgesic drugs including opioids (i.e., routine use of oral analgesics 5 or more times per week for greater than 3 weeks within the past 2 years);
* Alcoholism or drug abuse within 2 years prior to the Screening Visit or routine consumption of 3 or more alcohol containing beverages per day; Alcohol containing beverages are defined as one beer (5%), one glass of wine (11%) and one shot (40%) hard liquor;
* Surgeon's trauma rating of severe following surgery;
* Unwilling or unable to comply with all requirements outlined in the protocol;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Cooper SA, Desjardins PJ, Bertoch T, Paredes-Diaz A, Troullos E, Tajaddini A, Centofanti R, An R, Morella D. Analgesic efficacy of naproxen sodium versus hydrocodone/acetaminophen in acute postsurgical dental pain: a randomized, double-blind, placebo-controlled trial. Postgrad Med. 2022 Jun;134(5):463-470. doi: 10.1080/00325481.2021.2008180. Epub 2021 Dec 8. PMID 34878953
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at one center in the US between 12-MAR-2020 (first participant first visit) and 05-OCT-2020 (last participant last visit).
Pre-assignment Details: Overall, 221 participants were randomized into this post-operative dental pain study; 90 participants received naproxen sodium treatment, 87 participants received hydrocodone/APAP (acetaminophen) treatment, and 44 participants received placebo.
Groups:
- Naproxen Sodium: Participants received a single dose of naproxen sodium tablets 440 mg (220 mg × 2 tablets) after surgical teeth extractions
- Hydrocodone / APAP: Participants received a single dose of hydrocodone/acetaminophen tablets 10/650 mg (5/325 mg × 2 tablets) after surgical teeth extractions
- Placebo: Participants received a single dose of matching placebo tablets (2 tablets) after surgical teeth extractions
Period: Overall Study
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Started | 90 | 87 | 44
Completed | 85 | 84 | 42
Not Completed | 5 | 3 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: included all subjects who were randomized and received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo | Total
Number analyzed (Participants) | 90 | 87 | 44 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.3 (1.62) | 19.3 (1.69) | 19.3 (2.00) | 19.3 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 42 | 20 | 112
  Male | 40 | 45 | 24 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 18 | 6 | 42
  Not Hispanic or Latino | 72 | 69 | 38 | 179
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline pain intensity [Count of Participants; unit: Participants]
  Moderate | 34 | 36 | 17 | 87
  Severe | 56 | 51 | 27 | 134

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference Over 12 Hours (SPID 0-12)
Description: Pain intensity is measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each post dose time point, pain intensity difference (PID) is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. Sum of Pain Intensity Differences (SPIDs) was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID over 12 hours ranges from -120 to 120. A higher value indicates a better pain reduction.
Time Frame: Up to 12 hours postdose
Population: PP Population: all subjects in safety population who provided at least one pain assessment after the first dose of study drug and did not have any major protocol violations and completed the 12-hour assessments.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale*hours
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 86 | 83 | 43
Scores on a scale*hours | 53.20 (3.09) | 38.39 (3.14) | 13.57 (4.35)
Statistical Analysis 1: Comparison: Naproxen Sodium vs Hydrocodone / APAP; Test type: Superiority; p = 0.001, ANCOVA — All p-values were presented using two-sided test with alpha 0.05 and were considered statistically significant; LS Mean Difference = 14.81, 95% CI 2-sided [6.10 to 23.51]
Statistical Analysis 2: Comparison: Naproxen Sodium vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — All p-values were presented using two-sided test with alpha 0.05 and were considered statistically significant; LS Mean Difference = 39.63, 95% CI 2-sided [29.08 to 50.18]
Statistical Analysis 3: Comparison: Hydrocodone / APAP vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — All p-values were presented using two-sided test with alpha 0.05 and were considered statistically significant; LS Mean Difference = 24.82, 95% CI 2-sided [14.26 to 35.39]

2. Secondary Outcome: Total Pain Relief Over 12 Hours (TOTPAR 0-12)
Description: Pain relief is measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = A little relief, 2 = Some relief, 3 = A lot of relief, 4 = Complete relief). Total Pain Relief is calculated as the area under the curve of pain relief score over time for the given time period by multiplying the pain relief score at each time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. TOTPAR over 12 hours ranges from 0 to 48, a higher value indicates more pain relief.
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale*hours
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 86 | 83 | 43
Scores on a scale*hours | 28.41 (1.36) | 21.31 (1.39) | 10.63 (1.92)

3. Secondary Outcome: Total Pain Relief Over 6 Hours (TOTPAR 0-6)
Description: Pain relief is measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = A little relief, 2 = Some relief, 3 = A lot of relief, 4 = Complete relief). Total Pain Relief is calculated as the area under the curve of pain relief score over time for the given time period by multiplying the pain relief score at each time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. TOTPAR over 6 hours ranges from 0 to 24, a higher value indicates more pain relief.
Time Frame: Up to 6 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale*hours
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 86 | 83 | 43
Scores on a scale*hours | 14.53 (0.61) | 12.69 (0.62) | 5.14 (0.87)

4. Secondary Outcome: Sum of Pain Intensity Difference Over 6 Hours (SPID 0-6)
Description: Pain intensity is measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each post dose time point, pain intensity difference (PID) is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. Sum of Pain Intensity Differences (SPIDs) was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID over 6 hours ranges from -60 to 60. A higher value indicates a better pain reduction.
Time Frame: Up to 6 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale*hours
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 86 | 83 | 43
Scores on a scale*hours | 28.41 (1.46) | 24.35 (1.48) | 6.23 (2.05)

5. Secondary Outcome: Number of Participants Required or Did Not Reqiure Rescue Pain Medication
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 86 | 83 | 43
Participants
  Number of participants required rescue pain medication | 18 | 43 | 29
  Number of participants did not require any rescue pain medication | 68 | 40 | 14

6. Secondary Outcome: Amount of Rescue Medication
Description: To quantify the use of opioid analgesics in treatment of post-operative dental pain, the amount of rescue medications (opioids) was converted to a standard unit, which was Morphine Milligram Equivalent (MME) using below formula:
  MME/Day = Strength per Unit × (Number of units / Days supply) × MME conversion factor
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalent (MME)
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 18 | 43 | 29
Morphine Milligram Equivalent (MME) | 7.8 (3.08) | 9.3 (4.02) | 10.5 (4.50)

7. Secondary Outcome: Time to First Use of Rescue Medication
Description: If a subject did not take the rescue medication during the treatment period, (s)he was censored at the time of last assessment.
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 86 | 83 | 43
Hours | NA [NA to NA] — NA = not estimable due to insufficient number of participants with events. | 10.42 [8.27 to NA] — NA = not estimable due to insufficient number of participants with events. | 2.57 [1.83 to 7.60]

8. Secondary Outcome: Duration of Pain at Least Half Gone Over 12 Hours
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 86 | 83 | 43
Hours | 8.87 (0.46) | 6.57 (0.46) | 3.31 (0.64)

9. Secondary Outcome: Duration of Pain at Least Half Gone Over 6 Hours
Time Frame: Up to 6 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Naproxen Sodium | Hydrocodone / APAP | Placebo
Number analyzed (Participants) | 86 | 83 | 43
Hours | 4.60 (0.22) | 4.08 (0.22) | 1.49 (0.31)

ADVERSE EVENTS:
Time Frame: From first dose of the study drug administration until end of study treatment, up to 1 day
Groups:
- Hydrocodone/APAP: Participants received a single dose of hydrocodone/acetaminophen tablets 10/650 mg (5/325 mg × 2 tablets) after surgical teeth extractions
Arm/Group | Naproxen Sodium | Hydrocodone/APAP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/87 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/87 | 0/44
Other Adverse Events (participants affected / at risk) | 2/90 | 33/87 | 11/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium (N=90) | Hydrocodone/APAP (N=87) | Placebo (N=44)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 30 (53) | 9 (16)
General disorders and administration site conditions (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (1) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT04307940/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT04307940/SAP_001.pdf